CLINICAL TRIAL: NCT05562674
Title: Impact of Veteran Voices & Visions Peer Support Groups on Social Integration for Veterans With SMI/Psychosis
Brief Title: Impact of VVV Group for Veterans With SMI
Acronym: VVV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4376-P
Record Dates: First submitted 2022-09-27; First posted 2022-10-03 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Psychotic Disorders; Veterans
MeSH Terms: conditions — Psychotic Disorders | interventions — Self-Help Groups

STUDY DESIGN:
Intervention Model Description: This is a single arm trial evaluating the feasibility and acceptability of the manualized protocol the investigators develop.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Veteran Voices & Visions (VVV) (Experimental): This is the experimental condition, testing the manual the investigators have developed.
  Interventions: Behavioral: Support group

INTERVENTIONS:
Behavioral: Support group — This is a group-based, peer specialist and clinician co-facilitated psychosocial intervention for Veterans with SMI, called "Veteran Voices and Visions" (VVV). VVV is an adaptation of a community-based support group model called the Hearing Voices (HV) approach. The approach facilitates group cohesion around and normalization of the common psychotic symptoms of SMI: hallucinations, delusions, and social isolation.

SUMMARY:
Veterans with Serious Mental Illness (SMI) struggle with social integration - participation in work, housing, and citizenship - due to symptoms, stigma, and psychosocial challenges. Despite considerable VA efforts to provide mental health care to Veterans with SMI, programs that promote social integration are lacking. Veterans with SMI are at especially high risk for poor social integration and suicidal ideation during the COVID-19 pandemic. This project addresses this need with a group-based, peer specialist (PS) co-facilitated psychosocial intervention for Veterans with SMI, called "Veteran Voices and Visions" (VVV). VVV targets Veterans with SMI who experience psychosis, a group particularly in need of support with social integration. Virtual VVV groups are co-led by VA mental health clinicians (MHCs) and PSs via online video conference. The approach facilitates group cohesion around and normalization of the common psychotic symptoms of SMI: hallucinations, delusions, and social isolation. This intervention has the potential to create and foster a supportive community that improves the social integration of participants by reducing their distress and self-stigma, and increasing self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* DSM 5 diagnoses of schizophrenia, schizoaffective disorder, bipolar with psychosis, depression with psychosis, unspecified psychosis

Exclusion Criteria:

* Substance-induced psychosis,
* clinically significant neurological disease,
* history of serious head injury with loss of consciousness > 1 hour.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
The Psychotic Symptoms Rating Scale (PSYRATS-AHS) | 12 weeks after the initiation of the intervention.
  PSYRATS-AHS is an 11-item scale which assesses the frequency, duration, severity, loudness, location, negative content, and controllability of voices, intensity of distress, and beliefs about origin of voices and disruptiveness. Range of score is 0-44. The investigators will be assessing for within-subject change. Any decrease in overall score is indicative of decreased distress.

CONTACTS AND LOCATIONS:
Overall Officials: Ippolytos A Kalofonos, MD PhD MPH, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will create de-identified, study-specific datasets that include all variables in a publication. Some loss of information might occur given the need to remove PHI. The PI will replace social security and medical station numbers with study-specific numbers. The PI will drop date of birth and replace age with age categories, in accordance with PHI requirements for people 85 years of age and older. Dates of service will be replaced with year dummies.
Time Frame: Datasets meeting VA standards for disclosure to the public will be made available within 1 year of publication.
Access Criteria: Prior to distribution, a local privacy officer will certify that all datasets contains no PHI. Final data sets will be maintained locally until enterprise-level resources become available for long-term storage and access. Guidance on request and distribution processes will be provided by ORD. Those requesting data will be asked to sign a Letter of Agreement.

DOCUMENTS (1):
  • Informed Consent Form (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT05562674/ICF_000.pdf